CLINICAL TRIAL: NCT06321809
Title: The Effect of Intensive Lifestyle Intervention Applied to Overweight and Obese Patients in Primary Care During the Pandemic Period: a Randomised Controlled Trial
Brief Title: Intensive Lifestyle Interventions to Overweight and Obese Patients in Primary Care
Status: Completed | Type: Observational
Sponsor: Duygu Ayhan Baser (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Duygu Ayhan Baser, Assoc Prof, Hacettepe University
Organization: Hacettepe University (Other)
Other Study IDs: HUTF-FM-DABDCO-01
Record Dates: First submitted 2024-03-04; First posted 2024-03-20 (Actual); Results first posted 2025-02-04 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Life Style; Lifestyle, Sedentary
Keywords: primary care; obesity; lifestyle changes
MeSH Terms: conditions — Obesity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intervention group: They were given a calorie-restricted diet and exercise plan by a dietician or physiotherapist at their first visit, and were followed up by telephone calls at weeks 2, 4, 6, 8 and 10 over 12 weeks.
  Interventions: Behavioral: intensive lifestyle
- Control-1 group: During the initial medical interview, the participants were given a calorie-restricted diet programme by a dietician and an exercise programme by a physiotherapist; they were followed up over 12 weeks with telephone calls at week 4.
  Interventions: Behavioral: intensive lifestyle
- Control-2 group: The participants were not provided with any programme, and the importance of weight loss was emphasised by the family physicians. Dietary and physical activity advice was given according to the recommendations in the Turkish Endocrine and Metabolism Association 2019 Obesity Diagnosis and Treatment Guide, and was followed up with phone calls at weeks 2, 4, 6, 8 and 10 over a 12-weeks.

INTERVENTIONS:
Behavioral: intensive lifestyle — INTENSIVE LIFESTYLE INTERVENTIONS
  Groups: Control-1 group; Intervention group

SUMMARY:
The goal of this clinical trial is to compare in the effect of different lifestyle interventions in overweight and obese participants. The main questions it aims to answer are:

* effect on anthropometric measurements
* effect on lipid profile
* effect on weight-related quality of life
* observe the differences between interventions The study participants were stratified into three groups: intervention, control-1, and control-2.
* Intervention group: They were given a calorie-restricted diet and exercise plan by a dietician or physiotherapist at their first visit, and were followed up by telephone calls at weeks 2, 4, 6, 8 and 10 over 12 weeks.
* Control-1 group: During the initial medical interview, the participants were given a calorie-restricted diet programme by a dietician and an exercise programme by a physiotherapist; they were followed up over 12 weeks with telephone calls at week 4.
* Control-2 group: The participants were not provided with any programme, and the importance of weight loss was emphasised by the family physicians. Dietary and physical activity advice was given according to the recommendations in the Turkish Endocrine and Metabolism Association 2019 Obesity Diagnosis and Treatment Guide, and was followed up with phone calls at weeks 2, 4, 6, 8 and 10 over a 12-weeks.

DETAILED DESCRIPTION:
With this study, it is aimed to evaluate the effect of intensive lifestyle intervention to be applied to patients and follow-ups made by telephone calls in order to protect overweight and obese patients who apply to primary health care services from obesity and complications of obesity in the pandemic process in which the number of applications to secondary and tertiary care decreased due to pandemic conditions and the number of applications to primary care increased, in addition to this, the susceptibility to obesity increased due to changing lifestyle behaviours with the effect of the pandemic; The aim of this study is to evaluate the effect of intensive lifestyle intervention and telephone follow-ups on body mass index, body composition, lipid profile, obesity-related quality of life and to evaluate different forms of intervention organised as intensive lifestyle intervention and increasing the frequency of follow-up.

ELIGIBILITY:
Inclusion Criteria:

Age 18-40 BMI ≥ 25 kg/m 2 Agreeing to participate in the study Not having a diagnosed chronic disease To be able to ambulate To be cooperative

Exclusion Criteria:

* Receiving medical treatment
* Secondary obesity (hypothyroidism, Cushing's disease, etc.)
* Chronic disease (cardiovascular diseases, pulmonary diseases, presence of diabetes mellitus, liver diseases, renal diseases)
* Having hyperlipidaemia under treatment
* Cancer
* Pregnancy or breastfeeding
* Psychiatric disorder
* Orthopaedic or neurological disease that may prevent walking
* Are currently taking weight loss medication or enrolled in another weight loss program
* Having previously undergone obesity surgery or having surgery planned during the study period

Ages: 18 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: The study's participants comprised of overweight and obese individuals who made applications to the Department of Family Medicine at XXX University's Faculty of Medicine. Detailed information regarding the study was provided to overweight and obese individuals who applied between the dates of 25th January 2022 and 31st October 2022 and consented to participate in said study.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Ayhan Baser, Assoc. Prof., Study Director — Hacettepe University; Dilara Canbay Ozdemir, M.D., Principal Investigator — Hacettepe University; İzzet Fidanci, Assoc. Prof., Principal Investigator — Hacettepe University; Arzu Demircioglu Karagoz, Principal Investigator — Hacettepe University; Merve Ozdemir, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study's participants comprised of individuals with overweight and obese who made applications between the dates of 25th January 2022 and 1st October 2022 to the Department of Family Medicine.
Pre-assignment Details: Sixteen participants were excluded from the study. Six participants were excluded due to having a BMI of less than 25 kg/m2. Two participants were excluded due to pregnancy or breastfeeding, and five participants were excluded due to having a chronic disease.
  Three participants were excluded due to their age, being either under 18 years old or over 40 years old.
Period: Overall Study
Arm/Group | Intervention Group | Control-1 Group | Control-2 Group
Started | 55 | 56 | 54
Completed | 51 | 51 | 51
Not Completed | 4 | 5 | 3

BASELINE CHARACTERISTICS:
Population: It is identical to the assignment in Participant Flow or information about how participants contribute units.In the single-blind trial, patients were assigned to groups based on the order of admission. Randomization was performed using the blocked randomization technique with six blocks determined.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control-1 Group | Control-2 Group | Total
Number analyzed (Participants) | 51 | 51 | 51 | 153
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 51 | 51 | 153
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 35 | 107
  Male | 13 | 17 | 16 | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body Mass Index (kg/m2) [Count of Participants; unit: Participants]
  Overweight (BMI greater than or equal to 25) | 13 | 23 | 27 | 63
  Obese (BMI greater than or equal to 30) | 38 | 28 | 24 | 90

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome
Description: Turkish version of the Impact of Weight on Quality of Life-Lite Version (IWQOL) scale was used. The scale has a minimum score of 0 and a maximum of 100. The scoring system is valid for both the scale subgroups and the scale total score. Based on the scale scoring, quality-of-life decreases as the score decreases.
Time Frame: 3 months
Population: All participants were analysed.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Intervention Group | Control-1 Group | Control-2 Group
Number analyzed (Participants) | 51 | 51 | 51
score on a scale
  Physical function (baseline) | 68.18 [0 to 93.18] | 68.18 [4.55 to 97.73] | 70.45 [9.09 to 100]
  Self-esteem (baseline) | 50 [0 to 100] | 57.14 [0 to 96.43] | 50 [0 to 100]
  Sexual life (baseline) | 75 [0 to 100] | 87.50 [0 to 100] | 81.25 [0 to 100]
  Public distress (baseline) | 90 [15 to 100] | 85 [10 to 100] | 85 [0 to 100]
  Work (baseline) | 75 [0 to 100] | 87.50 [0 to 100] | 87.50 [0 to 100]
  Total Score (baseline) | 63.79 [16.38 to 95.69] | 73.28 [28.45 to 93.97] | 69.83 [18.97 to 99.14]
  Physical function (3 months) | 79.54 [0 to 100] | 77.27 [22.73 to 100] | 84.09 [0 to 100]
  Self-esteem (3 months) | 75 [0 to 100] | 82.14 [0 to 100] | 60.71 [3.57 to 100]
  Sexual life (3 months) | 87.50 [0 to 100] | 93.75 [25 to 100] | 93.75 [0 to 100]
  Public distress (3 months) | 90 [0 to 100] | 95 [30 to 100] | 90 [0 to 100]
  Work (3 months) | 87.50 [0 to 100] | 87.50 [12.50 to 100] | 87.50 [0 to 100]
  Total Score (3 months) | 81.90 [0 to 100] | 82.76 [33.62 to 100] | 81.03 [24.14 to 100]
Statistical Analysis 1: Comparison: Intervention Group vs Control-1 Group; total scale score comparison; Test type: Superiority; p = 0.24, Wilcoxon (Mann-Whitney); A significance level of p<0.05 was used for all analyses
Statistical Analysis 2: Comparison: Intervention Group vs Control-2 Group; total scale score comparison; Test type: Superiority; p = 0.001, Wilcoxon (Mann-Whitney); A significance level of p<0.05 was used for all analyses
Statistical Analysis 3: Comparison: Control-1 Group vs Control-2 Group; total scale score comparison; Test type: Superiority; p = 0.03, Wilcoxon (Mann-Whitney); A significance level of p<0.05 was used for all analyses
Statistical Analysis 4: Comparison: Intervention Group vs Control-1 Group vs Control-2 Group; total scale score comparison; Test type: Superiority; p = 0.003, Kruskal-Wallis; A significance level of p<0.05 was used for all analyses

2. Secondary Outcome: Secondary
Description: Comparing the anthropometric measurements of the three groups at baseline and week 12.
Time Frame: 3 months
Population: All participants were analysed.
Measure: Median (Full Range); unit: kg
Arm/Group | Intervention Group | Control-1 Group | Control-2 Group
Number analyzed (Participants) | 51 | 51 | 51
kg
  Weight (kg) (Baseline) | 89.50 [66.10 to 125.80] | 84.50 [61.90 to 135] | 85.10 [64.20 to 108.40]
  Fat mass (kg) (Baseline) | 33.50 [13 to 63.60] | 28.70 [17.20 to 48.80] | 26.80 [11.30 to 51.50]
  Fat free mass (kg) (Baseline) | 52.80 [43.10 to 83.30] | 50 [41.70 to 89.20] | 53.40 [40.70 to 78.60]
  Weight (kg) (3 months) | 88 [65.60 to 128.60] | 79.90 [58.80 to 135] | 84 [62.30 to 108.40]
  Fat mass (kg) (3 months) | 31.10 [13 to 64.20] | 28.80 [11.40 to 47.50] | 25.20 [5 to 51.50]
  Fat free mass (kg)(3 months) | 51.90 [43.40 to 82] | 48.50 [37.10 to 89.20] | 53.80 [41.90 to 75.30]
Statistical Analysis 1: Comparison: Intervention Group vs Control-1 Group vs Control-2 Group; Weight comparison; Test type: Superiority; p = 0.08, Kruskal-Wallis; A significance level of p<0.05 was used for all analyses

3. Secondary Outcome: BMI (kg/m2)
Description: Comparing the BMI of the three groups at baseline and week 12.
Time Frame: 3 months
Population: All participants were analysed.
Measure: Median (Full Range); unit: kg/m2
Arm/Group | Intervention Group | Control-1 Group | Control-2 Group
Number analyzed (Participants) | 51 | 51 | 51
kg/m2
  BMI (kg/m2) (Baseline) | 31.50 [25 to 47.30] | 30.50 [25.30 to 43.20] | 29.70 [25 to 42.30]
  BMI (kg/m2) (3 months) | 30.60 [24.30 to 48.40] | 29.50 [23 to 42.80] | 29.20 [24.80 to 42.30]
Statistical Analysis 1: Comparison: Intervention Group vs Control-1 Group vs Control-2 Group; BMI Comparison; Test type: Superiority; p = 0.13, Kruskal-Wallis; A significance level of p<0.05 was used for all analyses

4. Secondary Outcome: Waist Circumference (cm)
Description: Comparing the Waist Circumference measurements of the three groups at baseline and week 12.
Time Frame: 3 months
Population: All participants were analysed.
Measure: Median (Full Range); unit: cm
Arm/Group | Intervention Group | Control-1 Group | Control-2 Group
Number analyzed (Participants) | 51 | 51 | 51
cm
  Waist circumference (cm) (Baseline) | 106 [85.50 to 140] | 101.50 [77 to 158] | 101 [86 to 132]
  Waist circumference (cm) (3 months) | 102 [80 to 141] | 100 [70 to 158] | 100 [80.80 to 132]
Statistical Analysis 1: Comparison: Intervention Group vs Control-1 Group vs Control-2 Group; Waist Circumference Comparison; Test type: Superiority; p = 0.63, Kruskal-Wallis; A significance level of p<0.05 was used for all analyses

5. Secondary Outcome: Lipid Profile
Description: Lipid profile of the three groups at baseline and week 12.
Time Frame: 3 months
Population: All participants were analysed.
Measure: Median (Full Range); unit: mg/dL
Arm/Group | Intervention Group | Control-1 Group | Control-2 Group
Number analyzed (Participants) | 51 | 51 | 51
mg/dL
  Triglyceride (Baseline) | 105 [35 to 375] | 110 [39 to 231] | 94 [50 to 335]
  Total cholesterol (Baseline) | 188 [141 to 266] | 193 [131 to 284] | 181 [99 to 315]
  LDL cholesterol (Baseline) | 121 [68 to 180] | 120 [71 to 181] | 126 [74 to 231]
  HDL cholesterol (Baseline) | 45 [30 to 84] | 50 [31 to 90] | 46 [28 to 69]
  Triglyceride (3 months) | 100 [36 to 503] | 98 [45 to 230] | 96 [49 to 657]
  Total cholesterol (3 months) | 189 [120 to 282] | 189 [111 to 256] | 173 [105 to 324]
  LDL cholesterol (3 months) | 128 [70 to 193] | 125 [81 to 174] | 129 [88 to 258]
  HDL cholesterol (3 months) | 50 [33 to 87] | 48 [31 to 88] | 48 [27 to 67]
Statistical Analysis 1: Comparison: Intervention Group vs Control-1 Group vs Control-2 Group; LDL Cholesterol Comparison; Test type: Superiority; p = 0.89, Kruskal-Wallis; A significance level of p<0.05 was used for all analyses

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored.
Arm/Group | Intervention Group | Control-1 Group | Control-2 Group
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Yet, the three-month follow-up might not sufficiently capture lifestyle intervention impacts. Challenges in reaching participants during telephone follow-ups led to exclusions, potentially influencing the study's completeness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT06321809/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/09/NCT06321809/ICF_001.pdf